CLINICAL TRIAL: NCT03710018
Title: Localisation of Tumor Bed and Its Impact on Dosimetry for Tumor Bed Boost Irradiation in Patients Treated With Breast Conserving Surgery Using Different Techniques
Brief Title: Impact of Tumor Bed Localisation on Dosimetry Boost Irradiation in Patients Undergoing Breast Conserving Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. Ashwini Budrukkar, Associate Professor, Radiation Oncology, Tata Memorial Centre
Other Study IDs: 1860
Record Dates: First submitted 2018-07-24; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Breast Carcinoma
Keywords: Breast conservative surgery, tumor bed irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A Patient who underwent open cavity BCS: Patients undergoing Open cavity Breast Conservative Surgery
- B Patient who underwent close cavity BCS: Patients undergoing Close cavity Breast Conservative Surgery
- C Patient who underwent oncoplasty: Patients undergoing oncoplasty for breast cancer

SUMMARY:
PRIMARY STUDY OBJECTIVES:

To evaluate dosimetric outcomes in tumor bed boost irradiation in patients undergoing breast conservative surgery using three different surgical techniques SECONDARY OBJECTIVES- Evaluation of cosmesis in patients prior to radiotherapy, at the time of completion of radiotherapy and 6 months post completion of radiotherapy STUDY DESIGN: Three arm, Prospective Observational Trial

TREATMENT REGIMEN:

Group A- Patients who underwent open cavity Breast Conservative surgery(BCS) Group B- Patients who underwent closed cavity BCS Group C- Patients who underwent oncoplasty All patients will first receive external beam Radiotherapy to the whole breast to a dose of 40 Grays /15#/3 weeks. The patients will then be planned for boost radiation to the tumor bed to a dose of 12.5 Grays/5#.

RECRUITMENT TARGET: 20 Patients The sample size has not been calculated as this is a pilot study. Twenty patients will be accrued for the purpose of this study

PRIMARY ENDPOINT

1. Dosimetric Measurement

   * Seroma cavity volume (ccs).
   * PTV volume (ccs).
   * Ratio between the PTV volumes to the whole breast volume
   * Radiation Conformity Index (RCI)
   * Dose Homogeneity Index (DHI)
   * Ratio of dose received by 95% of PTV volume to the dose received by 5% of PTV volume
   * Dose received by several normal structures; normal ipsilateral breast tissue, contralateral breast, ipsilateral lung, contralateral lung, and heart
2. Cosmesis Measurement

   * prior to starting radiotherapy,
   * at the time of conclusion of radiotherapy
   * 6 months post completion of radiotherapy

DETAILED DESCRIPTION:
Introduction:

For patients with early stage invasive disease, surgery can either be a breast conserving resection of the primary tumor or a mastectomy. Several randomized prospective clinical trials have indicated that breast conserving surgery with whole breast radiation provides long term outcomes equivalent to those of mastectomy. The goal of breast conserving surgery is to remove the primary tumor with surgical margins that are free from invasive or in-situ disease. A secondary goal is to provide the best possible cosmetic outcome without retraction, nipple displacement, or excess volume loss from the procedure. For some women with larger breasts, oncoplastic surgery can be used in which local tissue rearrangements are performed at the time of surgical resection to maintain optimal breast aesthetics

Radiation is essential component of breast conserving therapy. The use of RT improved recurrence free, breast cancer specific survival and overall survival in both patients with negative and positive axillary lymph nodes in the most recent meta-analysis of Early Breast Cancer Trialists Collaborative Group(EBCTCG)5 which included trials begun before 2000.It included data from 42080 patients with breast cancer treated in 78 clinical trials that investigated loco regional treatments between 1952 and 1995.Among those patients were 7311 patients treated in 10 trials comparing radiation vs no radiation after breast conserving surgery and 9933 patients treated in 25 trials comparing radiation vs no radiation after modified radical mastectomy. In the trials that investigated radiation as a component of breast conserving therapy, radiation was shown to reduce the risk of local recurrence by two thirds and to improve the absolute 15 year overall survival rate by 6% (41% versus 35%).Similarly for patients with positive lymph nodes treated with modified radical mastectomy, radiation reduced the risk of loco-regional recurrence rate by 21% at 15 years(29% versus 8%), which was associated with a 5% decrease in the 15 year breast cancer mortality rate (60% versus 55%).A more recent update of the analyses continues to demonstrate loco-regional and survival advantages for radiation therapy

Even if surgical margins are negative after BCS, 30-40% risk of microscopic tumor cells in tumor bed. Most recurrences (65-80%) are located in vicinity of tumor bed as shown in EORTC6 trial and NSABP-06 trial. It is therefore important to ensure the tumor bed lies well inside the treatment volume encompassed by tangential fields to whole breast and subsequent tumor bed boost. There is also a pathological basis for giving boost to tumor bed-residual tumor foci have been reported in 1-2 cm in around 20-25% patients/ histopathological specimens.

The EORTC 22881-108827 trial studied the effect of addition of a boost dose on the primary tumor bed after lumpectomy in breast conserving treatment for breast cancer.It was found that 47% of local recurrences were in primary tumor bed, at 10 years, the cumulative incidence of local recurrence was 10.2% versus 6.2% for the 0 Grays and the 16 Grays boost groups (p< 0.0001).

The tumor beds of medially and laterally located tumors are particularly prone to under dosage if surface landmarks are used as fiduciary points for whole breast RT planning. It is therefore very important to localize the tumor bed even for whole breast RT planning.Clinical planning of tumor bed boost volume based on preoperative imaging, surgical note and breast scar position is very unreliable. Increasingly the breast scar is placed often some distance from the tumor for wire guided localisation biopsy or better cosmetic outcome. In addition the practice of oncoplastic surgery where breast tissue is re-positioned following wide excision to minimize the surgical deficit is becoming standard of care. In this situation the preoperative imaging bears very little final relation to tumor bed.

Computed tomography and ultra-sonography can use the seroma as a surrogate for tumor bed position, but there are limitations. First, the seroma is only clearly defined in only about quarter of patients. Second the seroma underestimates the tumor bed defined by implanted clips.

Uncertainty in localizing the tumor bed in medial or lateral tumors can be overcome by increasing the posterior field borders of whole breast tangents, but only at expense of increased morbidity of rib cage and lung, and potential mortality in women with left sided tumors. The heart is the most sensitive organ, a few Gy being associated with risk of heart disease and every effort needs to be made to exclude the organ from treatment volume. When localizing the tumor bed boost, increasing the clinical target volume is a crude way of avoiding geographical miss. This is particularly important in the era of oncoplastic surgery when the tumor bed may be well away from its primary location.

Accurate delineation of the target volume is of utmost importance while delivering tumour bed boost with external beam radiotherapy. Different institutions use different methods for delineation of the tumour bed.

Clinical history and patients' recollection of tumor position, clinical photographs, tattoos, surgical scar, mammography, surgical clips, ultra-sonography, Computerized tomography (CT) scan and Magnetic resonance imaging (MRI) are the commonly utilized techniques. Many a times, a combination of one or more of these techniques is considered while delineating the tumor bed boost.

Among all the randomized trials assessing role of radiotherapy boost, surgical clips were used in all patients for assessing boost volume only in the Budapest tria. It was hypothesized that increasing differences between local failure rates in whole breast radiotherapy (WBRT) arm versus WBRT+boost arm in Lyon trial (4.5% vs. 3.6%), EORTC trial (10.2% vs. 6.2%) and Budapest trial (15.5% vs. 6.7%) may well have been due to the different techniques of tumor bed delineation as the difference in boost doses between all these trials were not significantly different. Hence an accurate delineation of tumor bed is important as it may translate into improved local control rates.

Tumor bed localisation and open or closed cavity BCS: With superficial closure, only the superficial aspect of the cavity is closed, allowing the formation of a seroma to prevent deformation of the breast. A full-thickness closure consists of re-positioning of the surrounding breast tissue and suturing the deep and superficial layers, preventing the development of significant seroma. There is a paucity of data on the influence of surgical closure techniques on EB treatment planning. It can be hypothesized that superficial closure may lead to a better-delineated cavity as a well-visualized seroma has been shown to decrease inter observer variations nevertheless, it may also lead to a larger treatment volume and greater late toxicity effects. However, with full-thickness closure, the surgical clips may be displaced with the approximation of the surrounding breast tissue and not correlate with the true extend of the cavity. In a recently published single institutional experience,Shaikh . did not find statistically significant difference in mean cavity visualization scoring (CVS) or normal tissue dosimetric endpoints between 29 patients who underwent superficial closure and sixteen patients who underwent full-thickness closure. A higher percentage of patients who underwent superficial closure had CVS scores >2 (79% vs. 63%).

Neoplastic BCS techniques with parenchymal rearrangement present new challenges to the localisation of the tumor bed and therefore delivery of local boost radiotherapy. Although use of whole-breast radiation therapy (RT) is straight forward, difficulties in localization of the tumor bed for the local RT boost have not been investigated.Thus, in breast cancer patients who have undergone oncoplastic surgery, the tumor bed is frequently more extensive and possibly more relocated compared to original presentation. Placement of surgical clips after tumor resection and before oncoplastic reconstruction may be the most accurate method to localize the RT local boost field.

However, the boost fields defined on the basis of clinical details have been found to be erroneous in several studies. Hence, the dimensions as well as depth for tumor bed boost should be determined either by fluoroscopic or CT combined with surgical clips, or an ultrasound. The most common prescription isodose for electron boost delivery is 90-95% isodose. But, in an organ such as breast with multiple edges and curvatures in different axes, the prescription isodose may not cover the whole target volume uniformly. This problem is commonly seen when tumors are located at areas where there is a sudden change in the depths like inflammatory and axillary folds. The depths of soft tissue vary greatly in these areas and uniform energy electron beam may either underdose the tumor bed, or deliver higher dose to underlying normal structures. The electrons have limited role in patients with large breasts, tumors situated at a depth i.e. closer to heart (on left) and lungs and in folds. CT based planning in three dimensions may help to determine the dose distributions accurately and help in choosing the optimal energy.

The margins to be given to tumor bed for defining boost field have also been discussed. Harrington et al have shown that a boost field marked on the basis of clinical data and background with a margin of 2 cm all around covers radio logical field with same margin in only 1/3rd (33%) of patients. Although Vicini et al. showed that a margin of 1 cm around the tumor covers microscopic disease adequately, in EORTC trial margins of 1.5 cm were given for microscopically completely excised tumors. Overall, a margin of 1.5-2 cm to the tumor bed has been reported to cover all sub-clinical disease in patients with clear microscopic margins.

Some institutions have practiced tumor bed boost by 4-6 MV photons. The practice of delivering boost by photons has declined after widespread availability of electrons due to higher penetration and increased doses to underlying critical structures. Photons can be used in patients with small tumor bed as late term sequel of electrons such as telangiectasia may not be acceptable to some patients treated with electrons.

Material and methods- Patients will be screened for the study at the time of radiotherapy simulation for External beam radiotherapy

The sample size has not been calculated as this is a pilot study.Twenty patients will be accrued for the purpose of this study. The patients will be divided into three groups:

Group A- Patients who underwent open cavity BCS Group B- Patients who underwent closed cavity BCS Group C- Patients who underwent oncoplasty Inclusion Criteria- All patients undergoing Breast Conservative Surgery (Open Cavity/Closed Cavity) or Oncoplasty will be eligible for this study.

Exclusion Criteria-1.Patients undergoing Neoadjuvant chemotherapy will not be eligible for the purpose of this study.

2.All patients undergoing Modified Radical Mastectomy will not be eligible for the purpose of this study Informed consent will be taken for all patients at the time of Radiotherapy simulation. All patients will first receive external beam Radiotherapy to the whole breast to a dose of 40 Grays /15#/3 weeks. The patients will then be planned for boost radiation to the tumor bed to a dose of 12.5 Grays/5#.

The combination of surgical clips with a treatment planning CT scan for the lumpectomy site for electron boost and to determine the appropriate energy will be used for tumor bed boost delineation For the boost planning CT scan a small thermocol wedge will be used, with a pillow under the shoulder to make the surface as flat as possible.

The pT size in HPR of lumpectomy plus a margin of 2 cm in all directions is the approximate size of the boost field. The margins of this field are marked on the skin with the center of scar as the center of the field and copper wire is placed on the markings.

5 mm slice thickness CT scan will be taken in the treatment position. After the scan acquisition the data will be transferred to the Varian Eclipse treatment planning system.

The post-operative cavity depicted on the CT images will be contoured section by section. All available images will be assigned a cavity visualization score (CVS) as per the British Columbia Cancer Agency Cavity visualization score 0-No visible seroma, 1-scar/shadow, 2-seroma identifiable but with significant (>30%) uncertainties, 3-seroma identifiable with minor (<30%) uncertainties, 4- seroma easily identifiable, generally homogeneous with some blurring of margin, 5-seroma clearly identifiable, homogeneous with sharp boundaries. The mean cavity visualization score will be determined for each group of patients.

The CTV will be generated by using a 15 mm uniform expansion from the lumpectomy cavity but limited by skin and chest wall. The CTV will be extended by an additional 10 mm uniform expansion to generate the PTV Treatment plans for tumor bed boost irradiation will be made using both electrons and photons with 3DCRT technique for each patient and comparison will be made for various dosimetric variables. The photon beam plan will only be generated for purposes of dosimetric study and will not be used for treatment of the patients The following dosimetric variables will be determined for each patient -seroma cavity volume (ccs). PTV volume (ccs).In addition the ratio between the PTV volumes to the whole breast volume will be determined. The Radiation Conformity Index (RCI) will be determined for both set of plans. It was first defined by Knoos et al and a revised definition appeared in ICRU 62 It is the ratio of volume of the PTV to the volume that receives 95% prescribed dose or higher (RCI= V PTV/ V 95%). The Dose Homogeneity Index (DHI) will be determined for both set of plans (DHI). It is ratio of dose received by 95% of PTV volume to the dose received by 5% of PTV volume (DHI= D≥95%(within PTV) / D≥5% (within PTV) ). The dose received by several normal structures will be determined for both set of plans-normal ipsilateral breast tissue (Whole breast volume- PTV volume), contralateral breast, ipsilateral lung, contralateral lung and heart The borders of the portal will be modified based on the position of the lumpectomy cavity/seroma of the scan and marked on the patient. The boost irradiation for all patients will be done using electrons. The energy of electrons required will be decided from the depth of the lumpectomy cavity.

In addition the cosmesis will be determined for all the patients prior to starting radiotherapy, at the time of conclusion of radiotherapy and 6 months post completion of radiotherapy. This will be done by using the criteria suggested by Harris et al

ELIGIBILITY:
Inclusion Criteria:

1.All patients undergoing Breast Conservative Surgery (Open Cavity/Closed Cavity) or Oncoplasty will be eligible for this study.

Exclusion Criteria:

1. Patients undergoing Neoadjuvant chemotherapy will not be eligible for the purpose of this study.
2. All patients undergoing Modified Radical Mastectomy will not be eligible for the purpose of this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with breast cancer and eligible for the surgery
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Volume of PTV | at the time of radiation planning
  measured in cubic centimeter
PTV coverage by 95% isodose line | at the time of radiation planning
  measured in percent

SECONDARY OUTCOMES:
Cosmesis | on day of radiotherapy simulation, at 4 weeks post radiotherapy simulation and at 6 month post radiotherapy simulation
  Cosmesis will be evaluated using the JCRT criteria suggested by Harris et al

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Budrukkar, MD, DNB, Principal Investigator — Associate Professor, Tata Memorial Center, Mumbai India
Locations (1):
- Tata Memorial Center, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03710018/Prot_SAP_000.pdf